CLINICAL TRIAL: NCT00252551
Title: Vertebral Osteosynthesis in Degenerative Lumbar Stenosis With Spondylolisthesis - CLEOS Study
Brief Title: Vertebral Osteosynthesis in Degenerative Lumbar Stenosis With Spondylolisthesis
Acronym: CLEOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0300201; PHRC0300201 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Spondylolisthesis
Keywords: spondylolisthesis, decompressive surgery, osteosynthesis
MeSH Terms: conditions — Spondylolisthesis | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): osteosynthesis
  Interventions: Procedure: Osteosynthesis
- 2 (Active Comparator): Simple surgery
  Interventions: Procedure: Simple surgery

INTERVENTIONS:
Procedure: Osteosynthesis
  Arms: 1
Procedure: Simple surgery — Surgery without device
  Arms: 2

SUMMARY:
Study to evaluate the superiority of the osteosynthesis associated with a decompressive surgery in comparison with a simple decompressive surgery in the treatment of lumbar degenerative stenosis with spondylolisthesis

DETAILED DESCRIPTION:
Randomized, comparative study on 152 patients with degenerative spondylolisthesis L4-L5 confirmed by radiography with radicular pain for whom the antalgic and anti-inflammatory treatment are not efficient for at least 3 months.

Patients randomized in 2 parallel groups (each group with 76 patients)

* one group with decompressive surgery + osteosynthesis
* one group with decompressive surgery Study duration : 18 months, including a selection visit, an inclusion with the surgical intervention, 3, 12, 18 months' follow up visits and a follow up call at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative spondylolisthesis L4-L5 confirmed by radiography with radicular pain for whom the antalgic and anti-inflammatory treatment are not efficient for at least 3 months;
* Patients who agree to take part in the study and to sign an Informed Consent Form

Exclusion Criteria:

* Contre-indications to surgery or to vertebral isolated fixation L4-L5
* Previous lumbar surgery
* Work accidents
* Psychiatric troubles that may interfere with the clinical evaluation
* Pregnant women or women who could be pregnant during the study
* Patient under special supervision or trusteeship
* Refusal to sign the Informed Consent Form
* No Public Health Insurance cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the superiority of the osteosynthesis associated with a decompressive surgery in comparison with a simple decompressive surgery in the treatment of lumbar degenerative stenosis with spondylisthesis | M3, M12, M18

SECONDARY OUTCOMES:
improvement of patients' Quality of Life (SF36) | M18
radiologic stability of spondylolisthesis | M18
safety of the used surgical procedures | M3, M12, M18

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Lagarrigue, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - University Hospital of Besançon - Neurosurgey department, Besançon
  - University Hospital of Caen - Neurosurgery department, Caen
  - University Hospital of Clermont Ferrand, Clermont-Ferrand
  - Clinique Rech - Neurosurgery centre, Montpellier
  - University Hospital of Nice - Neurosurgery department, Nice
  - University Hospital of Saint-Etienne - Neurosurgery department, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg
  - Toulouse University Hospital - Purpan - Neurosurgery department, Toulouse
  - Toulouse University Hospital - Rangueil- Neuro surgery department, Toulouse

REFERENCES:
- [Background] Caputy AJ, Luessenhop AJ. Long-term evaluation of decompressive surgery for degenerative lumbar stenosis. J Neurosurg. 1992 Nov;77(5):669-76. doi: 10.3171/jns.1992.77.5.0669. PMID 1403105
- [Background] Cherkin DC, Deyo RA, Loeser JD, Bush T, Waddell G. An international comparison of back surgery rates. Spine (Phila Pa 1976). 1994 Jun 1;19(11):1201-6. doi: 10.1097/00007632-199405310-00001. PMID 8073310
- [Background] Davis H. Increasing rates of cervical and lumbar spine surgery in the United States, 1979-1990. Spine (Phila Pa 1976). 1994 May 15;19(10):1117-23; discussion 1123-4. doi: 10.1097/00007632-199405001-00003. PMID 8059266
- [Background] Feffer HL, Wiesel SW, Cuckler JM, Rothman RH. Degenerative spondylolisthesis. To fuse or not to fuse. Spine (Phila Pa 1976). 1985 Apr;10(3):287-9. PMID 3992350
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Gibson JN, Grant IC, Waddell G. The Cochrane review of surgery for lumbar disc prolapse and degenerative lumbar spondylosis. Spine (Phila Pa 1976). 1999 Sep 1;24(17):1820-32. doi: 10.1097/00007632-199909010-00012. PMID 10488513